CLINICAL TRIAL: NCT03313206
Title: Phase II Multicentric Study: Efficacy Evaluation of Neoadjuvant Treatment Associated With Maintenance Therapy by Anti-PD1 Immunotherapy on Disease-free-survival (DFS) in Patients With Resectable Head and Neck Mucosal Melanoma
Brief Title: Neoadjuvant Treatment Associated With Maintenance Therapy by Anti-PD1 Immunotherapy in Patients With Resectable Head and Neck Mucosal Melanoma
Acronym: IMMUQ
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Gustave Roussy, Cancer Campus, Grand Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2017-001628-23; 2017/2558 (Other: CSET number)
Record Dates: First submitted 2017-10-13; First posted 2017-10-18 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Head and Neck Mucosal Melanomas
MeSH Terms: interventions — pembrolizumab; Surgical Procedures, Operative; lenvatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort A (Experimental): The cohort A (Pembrolizumab only) will be opened in a first study step. Anti-PD1 antibody will be used (pembrolizumab, Merck®) intravenously at a dose of 200 mg every 3 weeks (4 injections maximum over 12 weeks), monotherapy
  Interventions: Drug: Pembrolizumab; Procedure: Surgery; Radiation: IMRT
- Cohort B (Experimental): Up to 26 evaluable patients will be treated in the cohort B (Pembrolizumab with Lenvatinib) if they do not have any contraindication for receiving lenvatinib treatment, otherwise they will be treated in the cohort A if slots are available. In the cohort B, the neo-adjuvant anti-PD1 immunotherapy will be combined with orally lenvatinib at a daily dose of 20 mg for 6 weeks started on the day of the first anti-PD1 dose.
  Interventions: Drug: Pembrolizumab; Procedure: Surgery; Radiation: IMRT; Drug: Lenvatinib

INTERVENTIONS:
Drug: Pembrolizumab — Neo-adjuvant therapy :
  * Anti-PD1 antibody will be used (pembrolizumab, Merck®) intravenously at a dose of 200 mg every 3 weeks. The patient will receive 4 injections maximum over 12 weeks. According to the investigator's opinion, the 4th injection might be cancelled in order to perform surgery from week 10 and not after week 13.
  * Tumor response will be assessed 2 weeks after the last injection both clinically and radiologically (by CT-scan and MRI).
  Maintenance therapy by anti-PD1 antibody (pembrolizumab, Merck®) will be then used intravenously at a dose of 200 mg every 3 weeks for a maximum period of one year, starting one month after the end of radiotherapy.
Procedure: Surgery — Surgery will be performed (endoscopically if possible) 3 weeks after the last injection, at the earliest week 10 and at the latest at week 13 and will be completed by radiotherapy using IMRT technology according to the International and European Rhinologic Societies guidelines.
Radiation: IMRT — Surgery will be performed (endoscopically if possible) 3 weeks after the last injection, at the earliest week 10 and at the latest at week 13 and will be completed by radiotherapy using IMRT technology according to the International and European Rhinologic Societies guidelines.
Drug: Lenvatinib — up to 26 evaluable patients will be treated with pembrolizumab combined with orally lenvatinib at a daily dose of 20 mg for 6 weeks started on the day of the first anti-PD1 dose.
  Arms: Cohort B

SUMMARY:
The main objective will be to estimate the disease free survival (DFS) of patients with resectable head and neck mucosal melanomas treated by neo-adjuvant anti-PD1 (in combination or not with lenvatinib) followed by surgery, radiotherapy and maintenance immunotherapy in order to compare it to historical DFS results of this kind of patients treated by surgery and radiotherapy. Our primary end-point will be disease-free survival at 2 years

ELIGIBILITY:
Inclusion Criteria:

1. Be willing and able to provide written informed consent/assent for the trial.
2. Be >/= 18 years of age on day of signing informed consent.
3. Present with a resectable head and neck mucosal melanoma.
4. Be eligible for surgical treatment (without any contraindications).
5. Be eligible for adjuvant radiotherapy.
6. Have measurable disease based on RECIST 1.1.
7. Be willing to provide tissue from a newly obtained core or excisional biopsy of a tumor lesion. Newly-obtained is defined as a specimen obtained up to 6 weeks (42 days) prior to initiation of treatment on Day 1. Subjects for whom newly-obtained samples cannot be provided (e.g. inaccessible or subject safety concern) may submit an archived specimen only upon agreement from the Sponsor.
8. Have a performance status of 0 or 1 on the ECOG Performance Scale.
9. Demonstrate adequate organ function as defined in table 1, all screening labs should be performed within 10 days of treatment initiation.
10. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
11. Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 120 days after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year.
12. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 120 days after the last dose of study therapy.
13. Patient affiliated to a social security system or beneficiary of the same

    For the cohort B, patients must met the following additional criteria :
14. Not having any contraindication for lenvatinib treatment

Exclusion Criteria:

1. Is currently participating and receiving study therapy or has participated in a study of an investigational agent and received study therapy or used an investigational device within 4 weeks of the first dose of treatment.
2. Has a metastatic disease.
3. Has a non resectable melanoma.
4. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (except topical or inhaled steroids) or any other form of immunosuppressive therapy within 2 weeks prior to the first dose of trial treatment.
5. Has a known history of active TB (Bacillus Tuberculosis)
6. Hypersensitivity to pembrolizumab or any of its excipients.
7. Has had a prior anti-cancer monoclonal antibody (mAb) within 4 weeks prior to D1 of study treatment or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to agents administered more than 4 weeks earlier.
8. Has had prior chemotherapy, targeted small molecule therapy, or radiation therapy within 4 weeks or 5 half-life times (whatever the shorter) prior to study Day 1 or who has not recovered (i.e., ≤ Grade 1 or at baseline) from adverse events due to a previously administered agent.

   * Note: Subjects with ≤ Grade 2 neuropathy are an exception to this criterion and may qualify for the study.
   * Note: If subject received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
9. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin or squamous cell carcinoma of the skin that has undergone potentially curative therapy or in situ cervical cancer.
10. Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment. This exception does not include carcinomatous meningitis which is excluded regardless of clinical stability.
11. Has active autoimmune and/or immune mediated inflammatory disease that has required systemic treatment in the past 2 years (i.e. with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
12. Has known history of, or any evidence of active, non-infectious pneumonitis.
13. Has an active infection requiring systemic therapy.
14. Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or is not in the best interest of the subject to participate, in the opinion of the treating investigator.
15. Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial.
16. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 120 days after the last dose of trial treatment.
17. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD L2 agent.
18. Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies).
19. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
20. Has received a live vaccine within 30 days of planned start of study therapy. Note: Seasonal influenza vaccines for injection are generally inactivated flu vaccines and are allowed; however intranasal influenza vaccines (e.g., Flu-Mist®) are live attenuated vaccines, and are not allowed.
21. Major injuries and/or surgery within the past 4 weeks prior to start of study treatment with incomplete wound healing
22. Has a prior history of organ transplant including allogeneic stem cell transplant
23. Has a LVEF below the institutional (or local laboratory) normal range, as determined by multigated acquisition (MUGA) or echocardiogram (ECHO)
24. Has an uveal melanoma

    For the cohort B, patients must be excluded if one of the following additional criteria is met :
25. Uncontrolled blood pressure (Systolic BP>140 mmHg or diastolic BP >90 mmHg) in spite of an optimized regimen of antihypertensive medication
26. Electrolyte abnormalities that have not been corrected
27. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, unstable angina, myocardial infarction or stroke within 12 months of the first dose of study drug, or cardiac arrhythmia requiring medical treatment at Screening
28. Bleeding or thrombotic disorders or subjects at risk for severe hemorrhage. The degree of tumor invasion/infiltration of major blood vessels (e.g. carotid artery) should be considered because of the potential risk of severe hemorrhage associated with tumor shrinkage/necrosis following lenvatinib therapy
29. Subjects having > 1+ proteinuria on urine dipstick testing unless a 24-hour urine collection for quantitative assessment indicates that the urine protein is <1 g/24 hours.
30. Subjects who have not recovered adequately from any toxicity from other anti- cancer treatment regimens and/or complications from major surgery prior to starting therapy. Withhold lenvatinib for at least 1 week prior to elective surgery. Do not administer for at least 2 weeks following major surgery and until adequate wound healing.
31. The participant has severe hypersensitivity (≥Grade 3) to lenvatinib and/or any of its excipients.
32. Has presence of a gastrointestinal condition including malabsorption, gastrointestinal, anastomosis, or any other condition that might affect the absorption of lenvatinib.
33. Has a pre-existing Grade ≥3 gastrointestinal or non-gastrointestinal fistula.
34. Has clinically significant hemoptysis or significant tumor bleeding within 3 weeks prior to the first dose of study drug.
35. Prolongation of QTcF interval to >480 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-05-28 (Actual); Primary Completion 2027-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Antoine MOYA PLANA, MD, Study Chair — Gustave Roussy, Cancer Campus, Grand Paris
Locations (1):
- Gustave Roussy, Villejuif, Val De Marne, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Gorry C, McCullagh L, O'Donnell H, Barrett S, Schmitz S, Barry M, Curtin K, Beausang E, Barry R, Coyne I. Neoadjuvant treatment for stage III and IV cutaneous melanoma. Cochrane Database Syst Rev. 2023 Jan 17;1(1):CD012974. doi: 10.1002/14651858.CD012974.pub2. PMID 36648215